CLINICAL TRIAL: NCT02102256
Title: A Feasibility Study of the Placement, Use, and Safety of the Nucleus 24 Auditory Brainstem Implant in Non-Neurofibromatosis Type 2 (NF2) Pediatric Patients
Brief Title: A Safety Study of the Auditory Brainstem Implant for Pediatric Profoundly Deaf Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laurie Eisenberg (Other)
Collaborators: University of Southern California (Other); Children's Hospital Los Angeles (Other); Huntington Medical Research Institutes (Other)
Responsible Party: Sponsor-Investigator, Laurie Eisenberg, Professor of Research Otolaryngology, University of Southern California
Organization: University of Southern California (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: KSOM-ABI 001
Record Dates: First submitted 2014-03-19; First posted 2014-04-02 (Estimated); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Profound Bilateral Deafness Due to; Bilateral Cochlear Aplasia; Bilateral Cochlear Nerve Deficiency; Bilateral Cochlear Ossification Secondary to Meningitis
Keywords: deafness; congenital; pediatric; device
MeSH Terms: conditions — Deafness | interventions — Auditory Brain Stem Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): Device Implantation
  Interventions: Device: Auditory Brainstem Implant

INTERVENTIONS:
Device: Auditory Brainstem Implant
  Other Names: Cochlear Corporation Nucleus 24

SUMMARY:
Current treatment options for bilateral profoundly deaf children, diagnosed with inner ear anatomical abnormalities, are limited and, in the case of absent cochleas, non-existent. An auditory brainstem implant (ABI) places an electrode close to the auditory nucleus in the brainstem. Children aged 2 - 5 who are not candidates for a cochlear implant, or who did not demonstrate benefit from a cochlear implant, will be implanted with an ABI and followed for 1 year for safety and a total of 3 years for preliminary efficacy. This is a feasibility study to determine the safety of the ABI.

DETAILED DESCRIPTION:
The multichannel auditory brainstem implant (ABI) has now been used with some benefit in more than 1000 deaf patients worldwide who were not candidates for a cochlear implant (CI). For many years, the ABI was used primarily in adults deafened by Neurofibromatosis-Type 2 (NF2). During the past decade, ABI surgery has been safely performed on non-NF2 children outside of the United States, and results have shown great promise. The overall objective of this Phase I Clinical Trial grant is to evaluate safety in ten pediatric subjects who are not candidates for traditional cochlear implants due to cochlear nerve deficiency, cochlear aplasia, or cochlear ossification. These types of pathologies prevent normal transmission of auditory information between the cochlea and the brainstem. The University of Southern California, House Clinic, and Children's Hospital of Los Angeles are conducting a pediatric, non-NF2 ABI clinical with the Nucleus ABI device.

The Primary Aim is to describe the safety aspects of device implant surgery and 12-month use of an ABI in 10 pediatric patients (ages 2-6 years) with profound bilateral hearing loss not amenable to other treatments, such as hearing aids or cochlear implants. Surgical safety analysis is defined as no greater number of serious surgery-related adverse events than is commonly observed in non-NF2 adults undergoing craniotomy with or without an ABI and no more than four unexpected serious device-related adverse events for the 10 subjects during 12 months of follow-up. A Secondary Aim will determine whether or not the device provides patients with access to sound (thresholds of 50 dB HL) during a critical period for communication skills development. Efficacy is here defined as access to sound at a level and within the frequency range, known to be associated with speech.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral profound deafness due to cochlear aplasia, cochlear nerve deficiency, or ossification secondary to meningitis
* If previously received a cochlear implant, must demonstrate lack of benefit from that device

Exclusion Criteria:

* Medical contraindication to craniotomy/intracranial surgery
* Severe cognitive or developmental delays

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurie S. Eisenberg, PhD, Principal Investigator — Keck School of Medicine of USC; Eric Wilkinson, MD, Principal Investigator — Huntington Medical Research Institute
Locations (2):
- United States (2):
  - Keck School of Medicine of USC, Los Angeles, California
  - Children's Hospital Los Angeles, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fisher LM, Eisenberg LS, Krieger M, Wilkinson EP, Shannon RV; Los Angeles Pediatric ABI Team. Regulatory and funding strategies to develop a safety study of an auditory brainstem implant in young children who are deaf. Ther Innov Regul Sci. 2015 Sep;49(5):659-665. doi: 10.1177/2168479015599559. No abstract available. PMID 26366332
- [Result] Wilkinson EP, Eisenberg LS, Krieger MD, Schwartz MS, Winter M, Glater JL, Martinez AS, Fisher LM, Shannon RV; Los Angeles Pediatric ABI Team. Initial Results of a Safety and Feasibility Study of Auditory Brainstem Implantation in Congenitally Deaf Children. Otol Neurotol. 2017 Feb;38(2):212-220. doi: 10.1097/MAO.0000000000001287. PMID 27898605
- [Result] Fisher LM, Martinez AS, Richmond FJ, Krieger MD, Wilkinson EP, Eisenberg LS. Assessing the Benefit-Risk Profile for Pediatric Implantable Auditory Prostheses. Ther Innov Regul Sci. 2018 Sep;52(5):669-679. doi: 10.1177/2168479017741111. Epub 2017 Nov 29. PMID 29714549
- [Result] Eisenberg LS, Hammes Ganguly D, Martinez AS, Fisher LM, Winter ME, Glater JL, Schrader DK, Loggins J, Wilkinson EP; Los Angeles Pediatric ABI Team. Early Communication Development of Children with Auditory Brainstem Implants. J Deaf Stud Deaf Educ. 2018 Jul 1;23(3):249-260. doi: 10.1093/deafed/eny010. PMID 29718280

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 10 subjects enrolled, 4 subjects did not proceed to auditory brainstem implant surgery because (1) the parents chose not to proceed, and/or (2) the child did not meet one or more of the inclusion criteria.
Groups:
- Auditory Brainstem Implant: Visit # 1 2 3 4 5 6 7 8 9 10 11-12 Day 0 Day 1-4 Wk 1 Wk 4-6 M 1 M 3 M 6 M 9 M 12 Yr 2-3 Activity Screen Implant In-hospital Activate device Device Fitting/Evaluation Early Efficacy Informed consent X Medical History X Audiological tests X Psychological tests X Vital signs X X X X Physical examination X Chest x-ray, EKG X Vaccinations X CT and MRI X Laboratory tests X Neurotology exam X X X X EABR X X Soundfield Thresholds X X X X X X Monitor vital signs X X X X X X X Device Fitting ("Mapping") X X X X X X X IT-MAIS/MAIS X X X X X X X Adverse Events X X X X X X X X X X Communication Battery X X
Period: Overall Study
Arm/Group | Auditory Brainstem Implant
Started | 6
Auditory Brainstem Implant Surgery (Undergo auditory brainstem implant surgery) | 6
Completed | 5
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Device Implantation
  Auditory Brainstem Implant
Arm/Group | Experimental
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: Years] — age at time of surgery or enrollment into the study
  Years | 3 [2 to 5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint
Description: Surgical Safety The number of subjects successfully implanted.
Time Frame: 12-months post-device (auditory brainstem implant) successful activation
Population: Deaf children receiving the auditory brainstem implant
Measure: Count of Participants; unit: Participants
Arm/Group | Auditory Brainstem Implant
Number analyzed (Participants) | 6
Participants | 6

2. Secondary Outcome: Secondary Endpoint: Preliminary Efficacy
Description: Access to sound at a level (dB HL) and with the frequency range (500-4000Hz), known to be associated with speech.
Time Frame: 3 years post-device activation
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 6
Participants
  250 Hz | 5
  500 Hz | 5
  1000 Hz | 5
  2000 Hz | 5
  4000 Hz | 5

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=10)
CSF leak following surgery resolved with lumbar drain (Ear and labyrinth disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=10)
Vestibular effects during electricial stimulation. Resolved by deprogramming affected electrode. (Ear and labyrinth disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/56/NCT02102256/Prot_000.pdf